CLINICAL TRIAL: NCT04516902
Title: Effects of MDMA Co-administration on the Response to LSD in Healthy Subjects
Acronym: LSD-MDMA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BASEC 2020-01829
Record Dates: First submitted 2020-08-13; First posted 2020-08-18 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Healthy
MeSH Terms: interventions — Lysergic Acid Diethylamide; N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, 4-period cross-over design with four treatment conditions:
  1. 100 μg LSD+MDMA placebo
  2. LSD placebo +100 mg MDMA
  3. 100 μg LSD + 100 mg MDMA
  4. LSD placebo+ MDMA placebo
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 100 μg LSD + MDMA placebo (Experimental): 100 μg LSD + MDMA placebo
  Interventions: Drug: Lysergic Acid Diethylamide; Other: MDMA Placebo
- LSD placebo +100 mg MDMA (Experimental): LSD placebo +100 mg MDMA
  Interventions: Drug: 3,4-methylenedioxymethamphetamine; Other: LSD Placebo
- 100 μg LSD + 100 mg MDMA (Experimental): 100 μg LSD + 100 mg MDMA
  Interventions: Drug: Lysergic Acid Diethylamide; Drug: 3,4-methylenedioxymethamphetamine
- LSD placebo+ MDMA placebo (Placebo Comparator): LSD placebo+ MDMA placebo
  Interventions: Other: LSD Placebo; Other: MDMA Placebo

INTERVENTIONS:
Drug: Lysergic Acid Diethylamide — A moderate dose of 100 μg LSD will be administered.
  Other Names: LSD
  Arms: 100 μg LSD + 100 mg MDMA; 100 μg LSD + MDMA placebo
Drug: 3,4-methylenedioxymethamphetamine — A moderate dose of 100 mg MDMA will be administered.
  Other Names: MDMA
  Arms: 100 μg LSD + 100 mg MDMA; LSD placebo +100 mg MDMA
Other: LSD Placebo — Pure alcohol instead of an alcoholic solution containing LSD
  Arms: LSD placebo +100 mg MDMA; LSD placebo+ MDMA placebo
Other: MDMA Placebo — Mannitol capsules instead of capsules containing MDMA
  Arms: 100 μg LSD + MDMA placebo; LSD placebo+ MDMA placebo

SUMMARY:
The acute subjective effects of serotonin (5-HT)2A receptor stimulation with lysergic acid diethylamide (LSD) in humans are mostly positive. However, negative effects such as anxiety, paranoid thinking or loss of trust towards other people are common effects, depending on the dose administered, the personality traits of the person consuming it (set), or the environment in which LSD is taken (setting). Negative psychedelic effects may cause acute distress to the subject and acute anxiety has been linked to less favourable long-term outcomes in patients experimentally treated with LSD or similar substances for the treatment of depression. The 5-HT and oxytocin releaser 3,4-methylenedioxymethamphetamine (MDMA) reliably induces positive mood up to euphoria, comfort, empathy, and feelings of trust. If administered in combination with LSD, MDMA may increase positive subjective drug effects including positive mood, empathy, and trust and reduce negative emotions and anxiety associated with LSD and overall produce a more positive over negative experience. The present study will assess subjective and autonomic effects of LSD alone and in combination with MDMA.

DETAILED DESCRIPTION:
LSD is a so-called "classic" or serotonergic hallucinogen or psychedelic. Its psychedelic effects are mainly attributed to its potent partial serotonin (5-HT) 5-HT2A receptor agonism. The effects of LSD have been frequently investigated in the past in both healthy participants and patients. Several of these studies described robust and sustained effects of LSD in patients suffering from addiction, anxiety and depression. The acute subjective effects elicited by LSD are mostly positive in humans. However, psychedelic substances like LSD may also cause unpleasant subjective effects like negative thoughts, rumination, anxiety, panic, paranoia, loss of trust towards other people and perceived loss of control, depending on the dose of LSD used, the personality traits of the person consuming it (i.e. 'set'), the environment in which it is consumed (i.e. 'setting'), and other factors yet to be determined. Acute negative psychological effects are considered the main risk of psychedelic substance use in humans. Inducing an overall positive acute response to the psychedelic is critical because several studies showed that a more positive experience is predictive of a greater therapeutic long-term effect of the psychedelic. Therefore, there is a need for methods which are capable of reducing bad drug effects while enhancing good drug effects to optimize a psychedelic experience.

The present study uses 3,4-methylenedioxymethamphetamine (MDMA) as a pharmacological tool to optimize LSD's effects profile by inducing positive mood. MDMA is an amphetamine derivative which, unlike prototypical amphetamines, predominantly enhances serotonergic neurotransmission via release of 5-HT through the serotonin transporter (SERT). Furthermore, MDMA is known to trigger oxytocin release which may contribute to its effects to increase trust, prosociality, and enhanced empathy. The state of well-being induced by MDMA including increased activation and emotional excitation is known to be associated with a better response to psychedelics. Due to its psychological profile, MDMA could be a reliable pharmacological tool to serve as an optimizer of a psychedelic experience by inducing positive emotions.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 25 and 65 years old
2. Sufficient understanding of the German language
3. Understanding of procedures and risks associated with the study
4. Willing to adhere to the protocol and signing of the consent form
5. Willing to refrain from the consumption of illicit psychoactive substances during the study
6. Abstaining from xanthine-based liquids from the evenings prior to the study sessions and during the sessions
7. Willing not to operate heavy machinery within 48 h of substance administration
8. Willing to use double-barrier birth control throughout study participation
9. Body mass index between 18-29 kg/m2

Exclusion Criteria:

1. Chronic or acute medical condition
2. Current or previous major psychiatric disorder
3. Psychotic disorder or bipolar disorder in first-degree relatives
4. Hypertension (SBP>140/90 mmHg) or hypotension (SBP<85 mmHg)
5. Use of hallucinogenic substances (not including cannabis) more than 20 times or any time within the previous two months
6. Use of MDMA more than 20 times or any time within the previous two months
7. Pregnancy or currently breastfeeding
8. Participation in another clinical trial (currently or within the last 30 days)
9. Use of medication that may interfere with the effects of the study medication
10. Tobacco smoking (>10 cigarettes/day)
11. Consumption of alcoholic beverages (>20 drinks/week)

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Acute subjective effects I | 12 months
  Visual Analog Scales (VAS) assessing the intensity and duration of subjective effects on a scale from 0% - 100% with higher scores representing more intense effects
Acute subjective effects II | 12 months
  Adjective Mood Rating Scale (AMRS) assesses the occurrence and intensity of 60 moods on a 4-point Likert scale ranging from "not at all" to "extremely"
Acute subjective effects III | 12 months
  5 Dimensions of Altered States of Consciousness (5D-ASC) consisting of 94 items to be rated on a visual analog scale (0-100 mm), with higher values indicating stronger effects
Autonomic effects I | 12 months
  Assessed 18 times on each study day via systolic and diastolic blood pressure
Autonomic effects II | 12 months
  Assessed 18 times on each study day via heart rate
Autonomic effects III | 12 months
  Assessed 18 times on each study day via tympanic body temperature

SECONDARY OUTCOMES:
Plasma levels of LSD | 12 months
  Assessed 18 times on each study day via blood samples
Plasma levels of MDMA | 12 months
  Assessed 18 times on each study day via blood samples
Plasma levels of blood-derived neurotrophic factor (BDNF) | 12 months
  Assessed 21 times on each study day via blood samples
Plasma levels of oxytocin | 12 months
  Assessed 4 times on each study day via blood samples
Psychological Insight Questionnaire | 12 months
  Assesses the degree of psychological insight caused by a psychedelic experience through 14-items to be answered on a 6-point Likert scale ranging from 0 ("not at all") to 5 ("extremely")
States of Consciousness Questionnaire | 12 months
  Assesses the emergence and intensity of phenomenons occurring in altered states of consciousness on a 6-point Likert scale ranging from 0 ("not at all") to 5 ("extremely")
Spiritual Realms Questionnaire | 12 months
  Assesses the spiritual phenomenons elicited by psychedelic substances through 11 main questions to be answered on a total of 65 sub-ordered 100mm visual analog scales
Effect moderation through personality traits I | Baseline
  Assessed via NEO-Five-Factor-Inventory (NEO-FFI)
Effect moderation through personality traits II | Baseline
  Assessed via Freiburger Personality Inventory (FPI)
Effect moderation through personality traits III | Baseline
  Assessed via Saarbrücker Personality Questionnaire (SPF)
Effect moderation through personality trait IV | Baseline
  Assessed via HEXACO personality inventory
Effect moderation through personality trait V | Baseline
  Assessed via Defense Style Questionnaire (DSQ-40)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, Prof. Dr. MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Clinical Trial Unit, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Straumann I, Ley L, Holze F, Becker AM, Klaiber A, Wey K, Duthaler U, Varghese N, Eckert A, Liechti ME. Acute effects of MDMA and LSD co-administration in a double-blind placebo-controlled study in healthy participants. Neuropsychopharmacology. 2023 Dec;48(13):1840-1848. doi: 10.1038/s41386-023-01609-0. Epub 2023 May 31. PMID 37258715